CLINICAL TRIAL: NCT06260358
Title: Multidisciplinary Assesssment of Structured Report for Cervical Cancer Staging
Acronym: STRECC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6043
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — MRI examinations will be performed on 1.5T or 3T scanners, with protocol according to ESUR guidelines.The contextual structured report will be generated by the investigators in consensus.
  In every centre, one report (structured or narrative) will be generated from various radiologists experienced in gynaecologic imaging during clinical practice. Two radiologists in consensus, will develop the second version (narrative or structured report).

SUMMARY:
This study aims to validate a structured report for cervical cancer anchored to the FIGO staging system. A structured report is hypothesized to aid in uniformly applying FIGO staging, reducing staging discrepancies and improving patient care and outcomes.

Furthermore, we believe that the participation of the clinicians will improve the quality of the report to minimize the need for multidisciplinary team discussion

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Overt biopsy-proven diagnosis of cervical cancer, at any stage;
* Signed written informed consent to personal data treatment for research purposes

Exclusion Criteria:

* Age <18 years old;
* Uncertain diagnosis of cervical cancer;
* MRI scan not according the standard acquisition protocol (ESUR guidelines);
* Patients candidate to non-standard treatments;
* Refusal to sign the written informed consent to personal data treatment for research purposes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven cervical cancer (any FIGO stage) undergoing staging MRI afferent to the participating centers satisfying the following inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a contextual structured report | 1 year
  Primary endpoint of the study is to assess referring physicians' (gynecologists and radiation oncologists) overall satisfaction rate with structured reports for staging MRI of patients with cervical cancer, in terms of overall response rate ≥4 at the first 5 items (i.e., an overall score ≥20)

SECONDARY OUTCOMES:
Satisfaction rate with narrative and structured report | 1 year
  To investigate the satisfaction rate of physicians between narrative and structured report
Comparison Single items response rate, on both narrative and structured reports | 1 year
  To compare Single items response rate (for items 6 to 12 of the questionnaire related to clinical information), on both narrative and structured reports.
Differences in the single 6-to-12 items response rate between structured and narrative reports. | 1 year
  To find differences in the single 6-to-12 items response rate between structured and narrative reports.

CONTACTS AND LOCATIONS:
Overall Officials: Evis Sala, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Advanced Radiology Center, Rome, Italy